CLINICAL TRIAL: NCT05802290
Title: A Single-Arm, Open-Label, Multicenter, Phase IIIb Clinical Trial With NIVolumab in Subjects With Recurrent or Metastatic Platinum-refrACTORy Squamous Cell Carcinoma of the Head and Neck (SCCHN) - NIVACTOR Study
Brief Title: NIVolumab in Subjects With Recurrent or Metastatic Platinum-refrACTORy SCCHN
Acronym: NIVACTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIVACTOR
Record Dates: First submitted 2021-01-18; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-05

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Injections

STUDY DESIGN:
Intervention Model Description: A Single-Arm, Open-Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab (Experimental): nivolumab monotherapy at 240mg flat dose as a 30-minute IV infusion on Day 1 of a treatment cycle every 2 weeks (14 days) until confirmed progression of disease, unacceptable toxicity, death or withdrawal of consent
  Interventions: Drug: Nivolumab 240 MG in 24 ML Injection

INTERVENTIONS:
Drug: Nivolumab 240 MG in 24 ML Injection — nivolumab monotherapy at 240mg flat dose as a 30-minute IV infusion on Day 1 of a treatment cycle every 2 weeks (14 days) until confirmed progression of disease, unacceptable toxicity, death or withdrawal of consent
  Other Names: Opdivo

SUMMARY:
Subjects will receive treatment with nivolumab monotherapy at 240mg flat dose as a 30 minute IV infusion on Day 1 of a treatment cycle every 2 weeks (14 days) until confirmed progression of disease, unacceptable toxicity, death or withdrawal of consent. This study is designed to better evaluate the safety profile of nivolumab in a large series of patients with Recurrent or Metastatic (R/M) Squamous Cell Carcinoma of the Head and Neck. The primary endpoint of this study is the incidence of high-grade (CTCAE v 4.03 Grade 3 or higher), treatment-related, select adverse events.

DETAILED DESCRIPTION:
This clinical trial has established head and neck squamous cell carcinoma as responsive to immunotherapy and nivolumab as a new potential SOC for these patients. As concern safety, high-grade (CTCAE v4.03 Grade 3 or higher), treatment-related, select adverse events occur with a low frequency in patients with Recurrent or Metastatic Platinum-refractory Squamous Cell Carcinoma of the Head and Neck (SCCHN) treated with nivolumab monotherapy. Nonetheless, this observation arises from patients treated in clinical trial and selected according to clear inclusion and exclusion criteria. Therefore they may not precisely reflect the clinical practice. Using a single large study is warranted in order to expand the safety database and to improve the knowledge on estimated incidence of uncommon, select, high-grade AEs.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent;
* Willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Males and Females, 18 years of age;
* Histologically confirmed recurrent or metastatic SCCHN (oral cavity, pharynx, larynx) not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy), p16 positive SCCHN of unknown primary;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Tumor progression or recurrence within 6 months of last dose of platinum therapy in the adjuvant (ie, with radiation after surgery), primary (ie, with radiation or prior to it or to surgery as induction chemotherapy), recurrent, or metastatic setting;
* Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria.
* Documentation of p16-positive or p16-negative disease to determine human papillomavirus (HPV) status of oropharyngeal cancer
* Tumor tissue (archival or fresh biopsy specimen) must be available;
* Patients with CNS metastases:

  * Patients are eligible if CNS metastases are treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, patients must be either off corticosteroids or on a stable or decreasing dose ≤ 10 mg daily prednisone (or equivalent) OR
  * Patients are eligible if they have previously untreated CNS metastases and are neurologically asymptomatic. In addition, patients must be either off corticosteroids or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent);
* Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration;
* Prior curative radiation therapy must have been completed at least 4 weeks prior to study drug administration. Prior focal palliative radiotherapy must have been completed at least 2 weeks before study drug administration
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test;
* Screening laboratory values must meet the following criteria (using CTCAE v4.03) and should be obtained within 14 days prior to the initial administration of study drug:

  * WBC ≥ 2000/μL
  * Neutrophils ≥1500/μL
  * Platelets ≥100 x103/μL
  * Hemoglobin ≥ 9.0 g/dL
  * Serum creatinine ≤ 1.5 x ULN o AST/ALT ≤ 3 x ULN
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
  * Calcium levels must be normalized and maintained within normal limits for study entry and on treatment. Medical management of calcium levels is permitted. Note: Normal calcium levels may be based on ionized calcium or adjusted for albumin.
  * Subjects with an initial magnesium < 0.5 mmol/L (1.2 mg/dL) may receive corrective magnesium supplementation but should continue to receive either prophylactic weekly infusion of magnesium and/or oral magnesium supplementation (eg, magnesium oxide) at the investigator's discretion.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post treatment completion;
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 halflives of study drug(s) plus 90 days (duration of sperm turnover) for a total of 31 weeks post treatment completion.

Exclusion Criteria:

* Patients with untreated, symptomatic CNS metastases are excluded;
* Histologically confirmed recurrent or metastatic carcinoma of the nasopharynx, p16 negative squamous cell carcinoma of unknown primary, and salivary gland or non-squamous histologies (eg, mucosal melanoma) are not allowed;
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results;
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti- CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways;
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast;
* Subjects with active, known or suspected autoimmune disease. Subjects with experienced GVH disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition or previous neck RT only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease;
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum-based therapy, are permitted to enroll.
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. Subjects who test positive for HCV antibody but negative for HCV ribonucleic acid are permitted to enroll;
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Any Grade 4 laboratory abnormalities;
* History of allergy to study drug components;
* History of severe hypersensitivity reaction to any monoclonal antibody;
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of high-grade (CTCAE v 4.03 Grade 3 or higher) treatment related AE | From baseline to 100 days after last study treatment
  To determine the incidence of high-grade (CTCAE v 4.03 Grade 3 or higher), treatment-related, select adverse events in patients with Recurrent or Metastatic Platinum-refractory Squamous Cell Carcinoma of the Head and Neck (SCCHN) treated with nivolumab monotherapy;

SECONDARY OUTCOMES:
Incidence of all high-grade (Grades 3-5), select adverse events; | From baseline to 100 days after last study treatment
  To determine the incidence and to characterise the outcome (duration of serious adverse events [SAE] treatment, dose of immune-modulating agents [ie, steroids] dose of agents used, time to event onset, and event resolution, and worst grade of event) of all high-grade (CTCAE v 4.03 Grade 3 or higher) adverse events
Overall Survival | At study end 2 years from last patient enrolled
  Defined as the time from first study treatment to death from any cause
Objective Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first (up to 24 moths)
  defined as the proportion of response-evaluable patients with a best overall response of CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, prof, Study Chair — Fondazione IRCCS Istituto Nazionale Tumori e Università di Milano
Locations (23):
- Italy (23):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Ospedale Bellaria, Bologna
  - IRCCS di Candiolo, Candiolo
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo - Cuneo (Cn) Oncoematologia, Cuneo
  - Az.Ospedaliera S.Croce e Carle, Cuneo
  - P.O. "Vito Fazzi", Lecce
  - Azienda USL Toscana Nord Ovest, Livorno
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Paolo, Milan
  - Istituto Tumori Napoli - Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale S.Chiara - A.O.U.P., Pisa
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Generale "S. Giovanni Calibita" Fatebenefratelli Isola Tiberina, Roma
  - Policlinico Universitario "Agostino Gemelli", Roma
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale S. Paolo, Savona
  - Ospedale San Paolo, Savona
  - AOU Città della Salute e della Scienza di Torino, Torino
  - ASST Vimercate, Vimercate